CLINICAL TRIAL: NCT03139708
Title: The Effect of Brimonidine on Intraocular Pressure When Dilating Routine Patients, Pressure Control and Pupil Effects
Brief Title: The Effect of Brimonidine on Intraocular Pressure When Dilating Routine Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00039213
Record Dates: First submitted 2016-10-05; First posted 2017-05-04 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Intraocular Pressure
Keywords: Mydriasis; Cycloplegics
MeSH Terms: conditions — Mydriasis | interventions — Brimonidine Tartrate; Phenylephrine; Tropicamide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The PI measuring pupil size will not know the subject assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Alphagan plus (Experimental): Alphagan plus group is one drop Brimonidine then, Tropicamide and Phenylephrine ophthalmic one drop,times one.
  Interventions: Drug: Alphagan; Drug: Phenylephrine; Drug: Tropicamide
- Tropicamide and Phenylephrine plus (Experimental): Tropicamide and Phenylephrine plus intervention is one drop of each then Brimonidine one drop, times one.
  Interventions: Drug: Alphagan; Drug: Phenylephrine; Drug: Tropicamide
- Tropicamide and Phenylephrine only (Active Comparator): Tropicamide and Phenylephrine only arm is given one drop of each times one.
  Interventions: Drug: Phenylephrine; Drug: Tropicamide

INTERVENTIONS:
Drug: Alphagan — Arm: Experimental: Alphagan plus Alphagan plus group is one drop Brimonidine then, Tropicamide and Phenylephrine ophthalmic one drop,times one.
  Arm: Experimental: Tropicamide and Phenylephrine plus Tropicamide and Phenylephrine plus intervention is one drop of each then Brimonidine one drop, times one.
  Other Names: Brimonidine
  Arms: Alphagan plus; Tropicamide and Phenylephrine plus
Drug: Phenylephrine — Arm: Experimental: Alphagan plus Alphagan plus group is one drop Brimonidine then, Tropicamide and Phenylephrine ophthalmic one drop,times one.
  Arm: Experimental: Tropicamide and Phenylephrine plus Tropicamide and Phenylephrine plus intervention is one drop of each then Brimonidine one drop, times one.
  Arm: Active Comparator: Tropicamide and Phenylephrine only Tropicamide and Phenylephrine only arm is given one drop of each times one.
Drug: Tropicamide — Arm: Experimental: Alphagan plus Alphagan plus group is one drop Brimonidine then, Tropicamide and Phenylephrine ophthalmic one drop,times one.
  Arm: Experimental: Tropicamide and Phenylephrine plus Tropicamide and Phenylephrine plus intervention is one drop of each then Brimonidine one drop, times one.
  Arm: Active Comparator: Tropicamide and Phenylephrine only Tropicamide and Phenylephrine only arm is given one drop of each times one.

SUMMARY:
This an interventional study looking at two different sequences of pre-operative eye drops, to determine which order is more effective in reducing intraocular pressure with pupil dilation.

DETAILED DESCRIPTION:
Twenty healthy participants will be separated into two groups of 10 volunteers each. In both groups, the participant's right eye will serve as a control with only Tropicamide/phenylephrine given. In one group of 10 participants the left eyes will receive Alphagan prior to Tropicamide/phenylephrine. In the other group of 10 eyes, the left eyes will have Tropicamide/phenylephrine administered prior to Alphagan. The investigator will observe the intraocular benefits of the addition of Alphagan over the Tropicamide/phenylephrine alone and determine if pre-treating is any better than post-treating. In addition, the investigator will monitor pupil response, as it is known that Alphagan may have some effect on the pupil dilation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy with no major medical conditions. Contact lens wear is ok but must be not worn on the day of the study

Exclusion Criteria:

* Diabetic, history of glaucoma
* history of iris trauma
* history of eye surgery except LASIK or Photorefractive keratectomy laser eye surgery
* Anisocoria
* pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in intraocular pressure from baseline to 15 min after last drop given, 30 min, 1 hour, and 4 hours. | 5 time points all occuring during one time visit: Baseline (pre drops), 15 min after last drop given, 30 min, 1 hour, and 4 hours.
  Baseline (pre drops), 15 min after last drop given, 30 min, 1 hour, and 4 hours.

SECONDARY OUTCOMES:
Change in pupil size pupil size from baseline to 15 min after last drop given, 30 min, 1 hour, and 4 hours. | 5 time points all occuring during one time visit: Baseline (pre drops), 15 min after last drop given, 30 min, 1 hour, and 4 hours.
  Baseline (pre drop), 15 min after last drop given, 30 min, 1 hour, and 4 hours. The investigator will measure the pupils under bright light conditions (photopic) and dim light conditions (scotopic)
Change in pupil's reaction to light from baseline to 15 min after last drop given,30 min, 1 hour, and 4 hours. | 5 time points all occuring during one time visit: Baseline (pre drops), 15 min after last drop given, 30 min, 1 hour, and 4 hours.
  Baseline (pre drop), 15 min after last drop given, 30 min, 1 hour, and 4 hours. Pupil reaction will be measure either as none, poor, or brisk.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Walter, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health Eye Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided